CLINICAL TRIAL: NCT07305857
Title: Comparison of the Effects of Target-Controlled Infusion Method and Manual Propofol Administration on Respiratory Function, Recovery, and Electroencephalogram in Endoscopic Submucosal Dissection Cases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, dilara gocmen, Dilara Göçmen, Marmara University Pendik Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2025/22/1301
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Endoscopic Submucosal Dissection; Target Controlled Infusion of Propofol; Endoscopy Unit; Respiratory Complications
Keywords: endoscopic submucosal dissection; target controlled infusion of propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manuel TIVA (Experimental): All patients will receive premedication with 0.03-0.05 mg/kg midazolam prior to the procedure. An ECG, SpO2, BIS, non-invasive blood pressure measurement, and Capnostream device nasal cannula will be applied to monitor EtCO2 by collecting exhaled air from the nose via a nasal cannula, and 5 L/min oxygen will be administered. All patients will receive 1-2 mcg/kg fentanyl intravenously.
  For patients in the Manual Group, anaesthesia maintenance will be performed with 1% propofol in accordance with routine anaesthesia practice. Bolus doses will be administered as needed during the procedure based on BIS, haemodynamics, and the patient's condition.
  Interventions: Procedure: manuel propofol and target controlled infusion propofol
- Group TCI (Experimental): All patients will receive premedication with 0.03-0.05 mg/kg midazolam prior to the procedure. An ECG, SpO2, BIS, non-invasive blood pressure measurement, and Capnostream device nasal cannula will be applied to monitor EtCO2 by collecting exhaled air from the nose via a nasal cannula, and 5 L/min oxygen will be administered. All patients will receive 1-2 mcg/kg fentanyl intravenously.
  For patients in the TCI group, a 1% propofol solution will be prepared in the perfusor, and the patient's height, weight, age, and gender will be entered into the device. The Schneider model, which calculates the dose based on pharmacokinetic models, will be used with a target plasma concentration of 0.5-3 µg/mL. Doses will be adjusted throughout the procedure based on the patient's BIS, haemodynamics, and condition.
  Interventions: Procedure: manuel propofol and target controlled infusion propofol

INTERVENTIONS:
Procedure: manuel propofol and target controlled infusion propofol — This study aims to compare the effects of manual TIVA and TCI propofol administration on recovery time, BIS, and respiratory parameters during ESD procedures performed in the endoscopy unit under sedation in the stomach or colon region. The findings will contribute to the safer and more effective planning of sedation procedures.

SUMMARY:
Endoscopic submucosal dissection (ESD) has become widely used as a minimally invasive alternative for the resection of early-stage gastrointestinal neoplasms. Due to the lengthy procedure time and intense pain caused by stretching, cutting, and dissecting the gastric wall during ESD, a deeper level of sedation is recommended compared to traditional endoscopic procedures (1). While ensuring adequate patient immobilisation during ESD, preserving respiratory function and rapid recovery are important clinical goals.

Total intravenous anaesthesia (TIVA) is an alternative method to inhalation anaesthesia, achieved through the combination of agents such as propofol and remifentanil. TIVA applications can be performed using manual or target-controlled infusion (TCI) systems. TCI systems aim to achieve and maintain the targeted plasma or effect site concentration based on pharmacokinetic models. These systems have been shown to provide advantages such as more stable depth of sedation during endoscopy, less haemodynamic fluctuation, and faster recovery (2-4).

Preserving spontaneous breathing is preferred during ESD procedures, which requires careful monitoring of respiration. The Capnostream® device records four variables (SpO₂, RR, non-invasive EtCO₂, heart rate) every 30 seconds via a nasal cannula and integrates them into a single, dimensionless value called the integrated pulmonary index (IPI). The IPI can range from 1 to 10, with 4 and below requiring intervention and 8 to 10 representing the normal range. Furthermore, the use of the bispectral index (BIS) enables objective monitoring of anaesthesia depth by analysing EEG waves and can increase the safety of the recovery process (5).

This study aims to compare the effects of manual TIVA and TCI applications on recovery time, BIS, and respiratory parameters during ESD procedures in the stomach or colon region performed under sedation in the endoscopy unit. The findings will contribute to the safer and more effective planning of sedation applications.

References;

1. Sasaki T, Tanabe S, Azuma M, Sato A, Naruke A, Ishido K, et al. Propofol sedation with bispectral index monitoring is useful for endoscopic submucosal dissection: a randomised prospective phase II clinical trial. Endoscopy. 2012 Jun;44(6):584-9.
2. Chang YT, Tsai TC, Hsu H, Chen YM, Chi KP, Peng SY. Sedation for gastrointestinal endoscopy with the application of target-controlled infusion. Turk J Gastroenterol Off J Turk Soc Gastroenterol. 2015 Sep;26(5):417-22.
3. Sarraj R, Theiler L, Vakilzadeh N, Krupka N, Wiest R. Propofol sedation in routine endoscopy: A case series comparing target controlled infusion vs manually controlled bolus concept. World J Gastrointest Endosc. 2024 Jan 16;16(1):11-7.
4. García Guzzo ME, Fernandez MS, Sanchez Novas D, Salgado SS, Terrasa SA, Domenech G, et al. Deep sedation using propofol target-controlled infusion for gastrointestinal endoscopic procedures: a retrospective cohort study. BMC Anaesthesiol. 10 August 2020;20(1):195.
5. Sandler NA, Hodges J, Sabino M. Assessment of recovery in patients undergoing intravenous conscious sedation using bispectral analysis. J Oral Maxillofac Surg Off J Am Assoc Oral Maxillofac Surg. 2001 Jun;59(6):603-11; discussion 611-612.
6. Ding Y, White PF. Simplified quality of anaesthesia scoring system. Anaesthesia. 1992 Oct;47(10):906-7.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old
* ASA (American Society of Anaesthesiologists) physical status class I-III
* Patients with indications for ESD
* BMI < 35 kg/m²
* Patients who are cooperative and can be monitored

Exclusion Criteria:

* Those with cardiac or pulmonary insufficiency,
* Those with neurological diseases,
* Those with severe hepatic or renal dysfunction,
* Those with psychiatric disorders that could affect their level of consciousness,
* Those with allergies or hypersensitivity to propofol, midazolam, and fentanyl, Patients who refuse to participate in the study will not be included in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
integrated pulmonary index value | while the procedure continues under anaesthesia
  Integrated pulmonary index values on the capnostream device
total apneic attack count | intraoperative time
  Number of apnoeic periods developing as a result of respiratory depression during the procedure

SECONDARY OUTCOMES:
total propofol dose (mg) | end of the case
  The amount of propofol used during the case shall be recorded in milligrams.
anaesthesia quality score(0-32) | intraoperative period
  The anaesthesia quality scoring scale, which assesses respiratory stabilisation and haemodynamic stability, will be used. The score obtained between 0 and 32 will be recorded.
post-operative recovery time | end of the case
  The time elapsed from the completion of the procedure until the patient opened their eyes and became cooperative.

IPD SHARING:
Plan to Share IPD: Undecided